CLINICAL TRIAL: NCT05900466
Title: Metformin as a Novel, Mechanistic Treatment of Fibromyalgia; a Proof of Concept RCT
Brief Title: Metformin for Fibromyalgia Symptoms (INFORM Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00160543; R21AR082574 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-06-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Fibromyalgia Syndrome
Keywords: FMS
MeSH Terms: conditions — Fibromyalgia | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: We will conduct a proof of concept pilot study, a single site, randomized, double-blinded, phase 2 clinical trial with 2 parallel dosing arms comparing the effects of placebo, and 500mg of once a day metformin on improving hyperalgesia and other symptoms in 72 patients with FMS.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1: Metformin Treatment (Active Comparator): 500 mg metformin ER tablets once daily in the morning with a glass of water for 8 weeks.
  Interventions: Drug: Metformin
- 2: Placebo (Placebo Comparator): Matching metformin ER placebo tablets once daily in the morning with a glass of water for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500 mg Metformin ER tablets once daily in the morning for 8 weeks
  Other Names: Glucophage XR (metformin hydrochloride); Glucophage (metformin hydrochloride)
  Arms: 1: Metformin Treatment
Drug: Placebo — Matching tablets once daily in the morning for 8 weeks
  Arms: 2: Placebo

SUMMARY:
The main purpose of the project is to evaluate the safety and efficacy of low dose metformin for improving symptoms associated with fibromyalgia syndrome (FMS) via modulating neuroinflammatory pathways. The investigators hypothesize that FMS patients in the low-dose metformin conditions will show greater improvement in FMS symptoms than those who are in the placebo group. Further, the investigators hypothesize that metformin will increase phosphorylated AMPK in peripheral immune cells of FMS patients and will decrease the transcription of mTORC1, NLRP3 inflammasome, and nociceptive cytokines interleukin 1beta and interleukin 18.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic pain condition that is debilitating to an estimated 10 million Americans and results in high utilization of medical resources with a cost of over $100 billion in health care and lost productivity each year. It is widely accepted that chronic widespread pain is a defining feature of FMS and that it is maintained by central sensitization. Accumulating evidence demonstrates that central sensitization is driven, at least in part, by neuroinflammation. Thus, molecules that ameliorate the causes of neuroinflammation are intriguing candidates to treat FMS symptoms. Current therapies are only partially effective in about 50% of patients. The development of a treatment approach with better efficacy is urgently needed.

The investigators propose to test the use of metformin for FMS. This drug is widely used as a first line treatment for type II diabetes. Metformin causes the phosphorylation of AMP-activated protein kinase (AMPK), which regulates key enzymes and transcription factors that modulate gene expression involved in metabolism and inflammation. Because AMPK acts as a master switch kinase, this target may prove particularly effective in treating the many diverse symptoms of FMS. Indeed, metformin treated hyperalgesia in preclinical models of neuropathic, inflammatory, spinal cord injury and diabetes-induced mechanical hyperalgesia and reduced symptoms of anxiety, depression and cognitive dysfunction. This is of significant relevance because these symptoms contribute greatly to FMS patient disability.

The investigators expect that this study will determine the effectiveness of metformin on pain and comorbidity FMS symptoms and delineate the role that AMPK and its downstream targets play on these phenotypes. The investigators anticipate that these results will demonstrate the efficacy of an intervention not currently used clinically to treat FMS. Understanding these pathways represents a critical step in the development of non-addictive pain treatments and holds enormous potential to reduce disability in the 10 million Americans with FMS.

ELIGIBILITY:
Inclusion Criteria:

* To be able to follow the protocol in English
* Fibromyalgia Syndrome: Participant must meet the American College of Rheumatology 2016 revised classification criteria for Fibromyalgia
* Ability to take oral medication and be willing to adhere to the metformin regimen (once daily)

Exclusion Criteria:

* Co-occurring progressive disease (self-report, physician-diagnosed)
* Diabetes
* Pregnancy or planning to be pregnant in the next year (all premenopausal participants will be tested)
* Having known cardiovascular, liver, kidney or pulmonary diseases (self-report, physician-diagnosed)
* Having known serious psychopathology (Clinician diagnoses of psychosis, organic mental disorder, or dissociative disorder, self-reported active suicidal intent, self-reported history of inpatient admission to a psychiatric ward in the past year, evidence or self-report of self-injurious behaviors in the past year, reported current or recent history (2years) of non-IV substance abuse, any history of recreational IV drug use)
* Having autoimmune disorder (e.g., rheumatoid arthritis) (self-report, physician-diagnosed)
* Having neuropathic pain (self-report, physician-diagnosed)
* Having pain associated with a terminal illness, acute pain, pain associated with specific organ damage (eg, stomach ulcer) (self-report, physician-diagnosed)
* Concurrent use of weight controlling medications (eg, Xenical)
* Requiring an interpreter to communicate
* Abnormal levels of creatinine, vitamin B12, or hepatic function panel
* eGFR of below 45mL/min/1.73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and efficacy of low-dose metformin in improving the symptoms associated with FMS | 12-14 weeks
  Safety will be measured by the Fibromyalgia Impact Questionnaire, Revised (FIQ-R score and will measure overall FMS severity. The numeric scale ranges from 0-10 with 0 being "low difficulty" (better outcome) and 10 being "high difficulty" (worse outcome).

SECONDARY OUTCOMES:
Examine changes in individual FMS symptoms - Pain Intensity | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of pain intensity (PROMIS Pain Intensity SF3a). The scale ranges from 0-10, 0 being "no pain" (better outcome) and 10 being "worst pain imaginable" (worse outcome).
Examine changes in individual FMS symptoms - Fatigue | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of fatigue (PROMIS Fatigue SF7a). The scale ranges from 1-5, 1 being "not at all" (better outcome) and 5 being "very much" (worse outcome).
Examine changes in individual FMS symptoms - Sleep Disturbance | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of sleep disturbance (PROMIS Sleep Disturbance SF8b). The scale ranges from 1-5, 1 being "very poor" or "not at all" (worse outcome) and 5 being "very good" or "very much" (better outcome).
Examine changes in individual FMS symptoms - Depression | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of depression (PROMIS Depression SF8b). The scale ranges from 1-5, 1 being "never" (better outcome) and 5 being "always" (worse outcome).
Examine changes in individual FMS symptoms - Anxiety | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of anxiety (PROMIS Anxiety SF7a). The scale ranges from 1-5, 1 being "never" (better outcome) and 5 being "always" (worse outcome).
Examine changes in individual FMS symptoms - Physical Function | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of physical functioning (PROMIS Physical Function SF10a). The scale ranges from 1-5, 1 being "unable to do" (worse outcome) and 5 being "without any difficulty" (better outcome).
Examine changes in individual FMS symptoms - Perceived Cognitive Function | 12-14 weeks
  Efficacy will be evaluated for a range of symptoms through the PROMIS Short Form measures of perceived cognitive functioning (title: Multiple Ability Self-Report Questionnaire (MASQ)). The scale ranges from 1-5 with 1 being "never" (better outcome) to 5 being "always" (worse outcome).
Examine changes in ecological momentary assessment (EMA) symptoms | 12-14 weeks
  EMA will allow us to evaluate symptom variations at home environment
Examine patient's global improvement impression | 12-14 weeks
  Global impression of improvement scale will be used to assess clinical global impression (CGI). Global impression of improvement scale is a 7-point scale. Scores range from 1 being the better outcome (i.e. "normal", "improved") and 7 being the worse outcome (i.e. "most severely ill", "very much worse").
Examine adherence | Week 4 and week 14
  Pill counts will provide us with a measure of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah; Norman Taylor, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States